CLINICAL TRIAL: NCT01231126
Title: Evaluation the Blood Loss in Pregnancies With Misoprostol-induced Labour
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maternidade Escola Assis Chateaubriand (Other)
Responsible Party: Paulo César Praciano de Sousa, Maternidade Escola Assis Chateaubriand
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 051/09
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2009-01

CONDITIONS: Pregnancy; Induced Labor
Keywords: Induced labor; Misoprostol; Postpartum blood; Erythrocyte indices; Vaginal delivery
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- spontaneous vaginal deliveries (Placebo Comparator)
  Interventions: Drug: Misoprostol
- elective caesarians (Placebo Comparator)
  Interventions: Drug: Misoprostol
- induced vaginal delivery by misoprostol (Experimental)
  Interventions: Drug: Misoprostol
- caesarians section with induction attempt (Experimental)
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — Procedures were taken for induced labor delivery with misoprostol 25mcg, by vaginal rout. The pills were administered each 6 hours in a maximum number of six.
  Other Names: Citotec

SUMMARY:
The purpose of this study is to evaluate the blood loss in induced vaginal delivery by misoprostol and caesarians section with induction attempt.

DETAILED DESCRIPTION:
Methods: it was a study achieved with 101 pregnant women with indication to induced delivery labor that were evaluated by the hemoglobin dosage pre and post delivery for estimate the blood loss at delivery. Patients were submitted to transabdominal obstetric ultrasound and basal cardiotocography. Procedures were taken for induced labor delivery with misoprostol 25mcg, by vaginal rout. The pills were administered each 6 hours in a maximum number of six. The control group was formed by 30 patients that began an spontaneously labor and 30 patients that achieved caesarians electively. The study of hemoglobin before and after delivery was evaluated through ANOVA to repeated measures, where it was verified the time effect (pre and post delivery) and the effect of the group (with and without use of misoprostol).

ELIGIBILITY:
Inclusion Criteria:

* Indication of early elective delivery by induction of labor (pre-eclampsia, HELLP syndrome, chronic hypertension, prolonged gestation, diabetes mellitus, gestational diabetes, heart disease, thyroid disease;
* pregnancy with living fetus;
* vertex cephalic presentation;
* estimated fetal weight by ultrasound > 2500g and <4000g;
* Amniotic fluid index (AFI)> 5 cm, except in cases of premature rupture of membranes in which AFI <5 cm would be allowed;
* cardiotocography (CTG) antepartum normal;
* Bishop Score less than or equal to 6;
* Determination of hemoglobin pre and post-partum.

Exclusion Criteria:

* Prior Cesarean section;
* previous uterine scar by myomectomy;
* Fetal presentation anomalous;
* Evidence of fetal abnormal (CTG, Ultrasound or Doppler);
* Fetal growth restriction;
* Gestation multiple;
* genital bleeding;
* tumors, malformations and / or ulceration in the region vulvoperineal and birth canal;
* No determination of hemoglobin pre-and post-partum;

Ages: 14 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 161 (Actual)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Vaginal delivery | 54 hours after the first pills
  Procedures were taken for induced labor delivery with misoprostol 25mcg, by vaginal rout. The pills were administered each 6 hours in a maximum number of six.

SECONDARY OUTCOMES:
blood loss | 24 hours after delivery
  To evaluate the blood loss in spontaneous vaginal deliveries and elective caesarians through the hemoglobin dosage pre and post delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo César Praciano de Sousa, Mestre, Principal Investigator — Maternidade Escola Assis Chateaubriand; Francisco Edson de Lucena Feitosa, Doutor, Study Director — Maternidade Escola Assis Chateaubriand
Locations (1):
- Maternidade-Escola Assis Chateaubriand, Fortaleza, Ceará, Brazil

REFERENCES:
- [Result] ElSedeek MSh, Awad EE, ElSebaey SM. Evaluation of postpartum blood loss after misoprostol-induced labour. BJOG. 2009 Feb;116(3):431-5. doi: 10.1111/j.1471-0528.2008.02054.x. PMID 19187376
- See also: site of Maternidade-Escola Assis Chateaubriand — http://www.meac.ufc.br